CLINICAL TRIAL: NCT04885569
Title: Feasibility Study of Culturally Adapted Cognitive Behavioral Therapy Based Integrated Motivational Interviewing and Mindfulness Intervention for Substance Use Disorder in Pakistan (CAMIAB)
Brief Title: Culturally Adapted Motivational Interviewing With CBT and Mindfulness Based Relapse Prevention for Substance Use Disorder in Pakistan (CAMIAB)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-CAMIAB-001
Record Dates: First submitted 2021-04-25; First posted 2021-05-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Substance Use Disorder (SUD)
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Motivational Interviewing with CBT (MICBT) (Experimental): Participants in this arm will receive a total of 12 weekly sessions of CBT based Motivational Interviewing over a period of 12 weeks.
  Interventions: Behavioral: Motivational interviewing with CBT (MICBT)
- Mindfulness based Relapse Prevention Group (MBRP) (Experimental): Participants in this arm will receive a total of 12 weekly sessions of mindfulness intervention over a period of 12 weeks.
  Interventions: Behavioral: Mindfulness based Relapse Prevention (MBRP)
- Integrated MICBT and MBRP Group (CAMIAB) (Experimental): This will be integrated MICBT plus MBRP intervention. Participants will receive a total of 12 weekly sessions of this integrated CAMIAB intervention.
  Interventions: Behavioral: CAMIAB
- Treatment as usual (TAU) (No Intervention): This will be routine care psychological treatment that they will be receiving.

INTERVENTIONS:
Behavioral: Motivational interviewing with CBT (MICBT) — The culturally adapted MICBT will include approaches of motivational interviewing and offer ways of managing difficulties from a cognitive behavioural formulation.
  Arms: Motivational Interviewing with CBT (MICBT)
Behavioral: Mindfulness based Relapse Prevention (MBRP) — MBRP will incorporate cognitive-behavioural skills (i.e., effective coping skills, self-efficacy, and recognizing common antecedents of relapse) with mindfulness-based practices to decrease the probability of relapse by increasing awareness and flexible responding in the presence of substance use triggers.
  Arms: Mindfulness based Relapse Prevention Group (MBRP)
Behavioral: CAMIAB — This will be integrated CBT based motivational interviewing plus mindfulness based relapse prevention intervention group.
  Arms: Integrated MICBT and MBRP Group (CAMIAB)

SUMMARY:
The study has both quantitative and qualitative components. The aim of study is to:

1. Culturally adapt and integrate the existing Motivational Interviewing with Cognitive Behavioral Therapy(MICBT) and Mindfulness based Relapse Prevention (MBRP) for people with Substance Use Disorder (SUD) in Pakistan
2. Test the feasibility and acceptability of the integrated intervention called CAMIAB ('CAMIAB' means success in Urdu) in a randomized control trial (RCT).

DETAILED DESCRIPTION:
This study aims to culturally adapt the existing Motivational Interviewing with CBT (MICBT) and integrate this with Mindfulness-Based Relapse Prevention (MBRP) intervention for people with SUD and to test the feasibility, and acceptability of the intervention in a randomized control trial (RCT). First phase will be cultural adaptation of intervention through focus groups and individual interviews with key stakeholders . Phase two will be to test integrated MICBT and MBRP on a small group of participants N=12.

Third phase will be a feasibility factorial randomized control trial with 260 participants with SUD (n=65). Participants will be recruited from primary care hospitals and drug rehabilitation centers in Karachi, Lahore, Rawalpindi, Hyderabad, and Peshawar Pakistan. Intervention will take place weekly over a period of 12 weeks. The intervention will consist of individual as well as group sessions. Assessments will be completed at baseline, after completion of intervention (12th week) and 24th week post randomization. All assessments will be administered by masked research assistants (RAs), not involved in delivering intervention sessions. The therapists delivering the intervention will be trained and will be provided ongoing supervisions by a senior therapist.

ELIGIBILITY:
Inclusion Criteria

* Participants with substance use disorder
* Meeting DSM-V criteria for substance use disorder
* Age 18 years and above
* Being able to understand spoken or written Urdu
* Have undergone through the process of detoxification before study intervention

Exclusion Criteria

• Any evidence of organic brain disease, clinically significant cooccurring medical illness or mental illness to the extent that can impede their ability to provide informed consent or engagement in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility measures | From baseline to 3rd month (at the end of intervention)
  Feasibility will be determined by recruitment rates, adherence rate and retention rates. The criterion for success of feasibility is to recruit >50% of eligible participants, adherence rate (number of home assignments completed; > 50%) and retention rate of 70%.
Acceptability measure | From baseline to 3rd month (at the end of intervention)
  Acceptability will be determined based on the number of sessions attended by participants and success criterion for intervention acceptability is mean attendance rate of at least 8 sessions.

SECONDARY OUTCOMES:
The Maudsley Addiction Profile | Change in problem scores from Baseline to 3rd Month and 6th month
  The Maudsley Addiction Profile is a brief, questionnaire that measures problems in four domains: substance use, health risk behaviour, physical and psychological health, and personal/social functions.
The Short Warwick-Edinburgh Mental Well-being Scale | Change in scores from baseline to 3rd Month and 6th month
  The Short Warwick-Edinburgh Mental Well-being Scale is a 7 items measure that will be used to measure mental wellbeing. It consists of 7 statements on a 5 point Likert scale. The minimum scale score is 7 and the maximum is 35. The high score indicates high mental wellbeing.
EuroQol-5 | Change in scores from baseline to 3rd Month and 6th month
  Quality of life will be measured using EuroQoL (EQ-5D) scale. This is a standardized instrument to measure health status and associated population utility weights. It measures five dimensions of health (mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression) at different levels that include "no problems, slight problems, moderate problems, severe problems, and unable to do/extreme".
Client service receipt inventory | Changes from baseline to 3rd Month and 6th month
  CSRI will be used to estimate the health and social services received.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Bashir Chaudhry, Prof., Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Pakistan Recovery Oasis, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asif M, Khoso AB, Husain MA, Shahzad S, Van Hout MC, Rafiq NU, Lane S, Chaudhry IB, Husain N. Culturally adapted motivational interviewing with cognitive behavior therapy and mindfulness-based relapse prevention for substance use disorder in Pakistan (CAMAIB): protocol for a feasibility factorial randomised controlled trial. Pilot Feasibility Stud. 2023 Apr 24;9(1):67. doi: 10.1186/s40814-023-01296-0. PMID 37095571